CLINICAL TRIAL: NCT01426165
Title: Effect of Magnesium Sulfate Infusion Rate on Magnesium Retention in Critically Ill Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with recruitment. PI decided to terminate study
Sponsor: CAMC Health System (Other)
Collaborators: Sarah & Pauline Maier Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Carol Morreale, Clinical Pharmacist Specialist - Emergency Medicine/Critical Care; Director, PGY2 Pharmacy Residency in Critical Care, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-10-2271
Record Dates: First submitted 2011-08-24; First posted 2011-08-31 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Primary Hypomagnesemia (Disorder)
Keywords: hypomagnesemia; magnesium; magnesium sulfate
MeSH Terms: conditions — Hypomagnesemia primary | interventions — Magnesium Sulfate; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium 8 grams over 4 hours (Experimental)
  Interventions: Drug: Magnesium Sulfate
- Magnesium 8 grams over 8 hours (Experimental)
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — 8 grams over 4 or 8 hours depending on randomization
  Other Names: magnesium

SUMMARY:
Hypomagnesemia (low magnesium) is an electrolyte imbalance commonly found in up to 65% of critically ill patients. Possible consequences of hypomagnesemia include neuromuscular and neurologic dysfunction, heart arrhythmias, and alterations in other electrolytes. Data has shown that critically ill patients with hypomagnesemia have a significantly higher mortality rate than patients with a normal magnesium level. The most simple and commonly used test to diagnose hypomagnesemia is a serum magnesium level. Based on the magnesium level and symptoms of hypomagnesemia, patients may be replaced with either oral or intravenous (IV) magnesium. When replacing magnesium via the IV route, approximately half of the dose is retained by the body while the remainder is excreted in the urine. The low retention rate is due to the slow uptake of magnesium by cells and decreased magnesium reabsorption by the kidneys in response to the delivery of a large concentration of magnesium. The purpose of this study is to determine whether an eight hour compared to a four hour infusion of IV magnesium sulfate results in a greater retention of the magnesium dose.

DETAILED DESCRIPTION:
Hypomagnesemia is a common electrolyte disturbance that affects up to 65% of intensive care unit (ICU) patients with normal renal function. Causes of hypomagnesemia are attributed to either gastrointestinal (secretory loss, impaired absorption or reabsorption, acute pancreatitis) or renal losses (alcohol, hypercalcemia, volume expansion, loop or thiazide diuretics, nephrotoxic medications, renal tubular dysfunction, inborn disorders). Consequences of magnesium deficiency are not benign and may include neuromuscular and neurologic dysfunction, cardiac arrhythmias and concomitant electrolyte abnormalities including hypokalemia and hypocalcemia. Hypomagnesemia has been associated with a significantly greater mortality rate in critically ill medical patients compared to normomagnesemic patients. In a study conducted by Rubeiz et al, 46% (17/37) of hypomagnesemic patients in the medical ICU died compared to 25% (37/147) of normomagnesemic patients (p < 0.05).

It can be difficult to assess patients for hypomagnesemia because of the unreliable relationship between serum and tissue magnesium levels. Approximately 1% of total body magnesium is found in the extracellular fluid while the remaining 99% is distributed among the bones, muscles, and soft tissues. Approximately 60% of serum magnesium is free ions; 33% is bound to proteins and 7% is complexed with anions. The most simple and commonly used test to diagnose hypomagnesemia is the total serum magnesium level which reflects free magnesium along with complexed and protein bound magnesium. The serum magnesium level, however, is not always accurate at detecting magnesium deficiency. Patients may appear to be normomagnesemic based on their serum magnesium level, yet have an underlying magnesium deficiency. Normal serum magnesium levels vary by laboratory. The normal range of values at Charleston Area Medical Center (CAMC) is 1.6-2.6 mg/dL.

Magnesium replacement depends on the clinical situation and manifestations. In critical conditions such as pre-eclampsia, arrhythmias, and tetany, large doses of IV magnesium are rapidly bolused and often followed by a continuous IV infusion. In asymptomatic patients, magnesium may be replaced by the oral or IV route depending on the clinical situation. The dose required to return patients to the normal magnesium range is variable and replacement may take several doses. Serum magnesium levels are primarily controlled by glomerular filtration and tubular reabsorption at the sites of the Loop of Henle and distal tubule. When faced with an increased filtered load of magnesium, the kidney is capable of increasing its excretion rate. Following intravenous (IV) administration, cellular magnesium uptake is slow and approximately 50% or more of the infused dose is lost due to increased excretion by the kidneys and decreased tubular reabsorption.

The investigators current practice in the Medical and Neuroscience ICUs at CAMC General Hospital is to order 8g of magnesium sulfate for replacement in patients with hypomagnesemia. When IV magnesium sulfate is ordered the pharmacy automatically sets the rate to run at 2g per hour unless otherwise specified. Often times the physician will specify for 8g to be infused over eight hours. The basis of using an extended infusion is that a slower magnesium infusion rate may increase magnesium retention by allowing a longer period of time for magnesium uptake by cells and by decreasing the magnesium load delivered to the kidneys at any given time. As far as the investigators are aware, there have been no studies completed to date that assess the rate of IV magnesium infusion on the magnesium retention rate.

ELIGIBILITY:
Inclusion Criteria:

Medicine ICU service patients

* > 18 years old with
* hypomagnesemia defined by a serum magnesium level < 2 mg/dL and the clinical decision by the rounding team to replace with parenteral magnesium sulfate
* must have an available IV line for magnesium infusion that may be used for up to 8 hours
* must have a Foley catheter

Exclusion Criteria:

* renal dysfunction defined by an estimated creatinine clearance (CrCl) < 30 mL/min or have had an average of < 0.5 mL/kg/hr of urine output over the previous 12 hours before the magnesium infusion is to begin
* Subjects must not have received a loop diuretic within the 12 hours prior to magnesium replacement and will further be excluded if they receive these medications during the magnesium replacement and urine collection time period
* Subjects with ostomies or acute diarrhea will be excluded due to the possibility of high gastrointestinal magnesium loss
* Subjects will be excluded if they have a physician order for magnesium sulfate to be infused over a specified time period
* If subjects are expected to be moved out of the ICU within the next 24 hours, they will not be considered for randomization due to potential lack of appropriate urine magnesium collection and follow up
* Each subject may only be enrolled in the study for one occurrence of hypomagnesemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Amount of urinary excretion of magnesium after an 8g magnesium sulfate infusion delivered over 4 hours versus 8 hours. | 24 hours

SECONDARY OUTCOMES:
Mean change in the serum magnesium level after an 8 gm magnesium sulfate infusion delivered over 4 hours and 8 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jack L DePriest, MD, Principal Investigator — WVU School of Medicine/Charleston Division
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

REFERENCES:
- [Background] Ryzen E, Wagers PW, Singer FR, Rude RK. Magnesium deficiency in a medical ICU population. Crit Care Med. 1985 Jan;13(1):19-21. doi: 10.1097/00003246-198501000-00006. PMID 3965244
- [Background] Epstein M, McGrath S, Law F. Proton-pump inhibitors and hypomagnesemic hypoparathyroidism. N Engl J Med. 2006 Oct 26;355(17):1834-6. doi: 10.1056/NEJMc066308. No abstract available. PMID 17065651
- [Background] Broeren MA, Geerdink EA, Vader HL, van den Wall Bake AW. Hypomagnesemia induced by several proton-pump inhibitors. Ann Intern Med. 2009 Nov 17;151(10):755-6. doi: 10.7326/0003-4819-151-10-200911170-00016. No abstract available. PMID 19920278
- [Background] al-Ghamdi SM, Cameron EC, Sutton RA. Magnesium deficiency: pathophysiologic and clinical overview. Am J Kidney Dis. 1994 Nov;24(5):737-52. doi: 10.1016/s0272-6386(12)80667-6. PMID 7977315
- [Background] Rubeiz GJ, Thill-Baharozian M, Hardie D, Carlson RW. Association of hypomagnesemia and mortality in acutely ill medical patients. Crit Care Med. 1993 Feb;21(2):203-9. doi: 10.1097/00003246-199302000-00010. PMID 8428470
- [Background] McLean RM. Magnesium and its therapeutic uses: a review. Am J Med. 1994 Jan;96(1):63-76. doi: 10.1016/0002-9343(94)90117-1. PMID 8304365
- [Background] Zaloga GP. Interpretation of the serum magnesium level. Chest. 1989 Feb;95(2):257-8. doi: 10.1378/chest.95.2.257. No abstract available. PMID 2914469
- [Background] CHESLEY LC, TEPPER I. Some effects of magnesium loading upon renal excretion of magnesium and certain other electrolytes. J Clin Invest. 1958 Oct;37(10):1362-72. doi: 10.1172/JCI103726. No abstract available. PMID 13575537
- [Background] BARKER ES, ELKINTON JR, CLARK JK. Studies of the renal excretion of magnesium in man. J Clin Invest. 1959 Oct;38(10 Pt 1-2):1733-45. doi: 10.1172/JCI103952. No abstract available. PMID 13796804
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Agus ZS. Hypomagnesemia. J Am Soc Nephrol. 1999 Jul;10(7):1616-22. doi: 10.1681/ASN.V1071616. No abstract available. PMID 10405219